CLINICAL TRIAL: NCT01868620
Title: Non-inferiority Trial of Iontophoretic Corneal Collagen Crosslinking (CXL) Compared to Standard Corneal Collagen Crosslinking in Progressive Keratoconus.
Acronym: IONTO-CXL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator decided to stop the trial due to a lack of inclusion.
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Sooft Italia (Industry); Centre de Référence National du Kératocône (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 030 03; HAO (Other: University Hospital of Toulouse)
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Progressive Keratoconus
Keywords: Progressive keratoconus; standard CXL; iontophoretic CXL; keratometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iontophoretic CXL (Experimental): The iontophoretic CXL involves a constant current source and two electrodes. The main electrode is a circular cup, with a surrounding annular suction ring to affix the device on the cornea during the procedure. The electrode itself is a stainless steel grid, placed into the cup at a minimal distance from the cornea. The reservoir is filled with riboflavin solution. The generator applies a constant current of 1mA for a preset period of 5 min. After the riboflavin administration by iontophoresis, the cornea is irradiated by a UVA light for 3mW/cm2 during 30 minutes.
  Interventions: Device: Iontophoretic CXL
- Standard CXL (Active Comparator): In the standard CXL, the epithelium is mechanically removed. Then, a solution of riboflavin is instilled each minute for 30 minutes. Corneas are irradiated by a UVA light for 3mW/cm2 during 30 minutes.
  Interventions: Device: Standard CXL

INTERVENTIONS:
Device: Iontophoretic CXL
  Arms: Iontophoretic CXL
Device: Standard CXL
  Arms: Standard CXL

SUMMARY:
The primary purpose of the protocol is to compare the current standard CXL with iontophoretic CXL to provide evidence in relation to the efficacy and safety in progressive keratoconus.

Corneal collagen crosslinking (CXL) is the first surgical procedure that appears to halt the progression of keratoconus. In the current standard CXL, the central corneal epithelium must be debrided to efficiently permeate the corneal stroma with riboflavin. The epithelium debridement can cause severe pain, infection and stromal haze. The study hypothesis is that iontophorese CXL is as effective as standard CXL to stabilize a progressive keratoconus.

DETAILED DESCRIPTION:
Keratoconus is a common bilateral progressive corneal ecstatic disease causing visual impairment by inducing irregular astigmatism and corneal opacities. This disorder typically begins during teenage years, progresses until the age of 30 to 40 years and, in severe forms, may need a corneal transplantation. CXL has changed the natural evolution of keratoconus. It creates links between collagen fibrils in order to rigidify the corneal stroma and slow down the progression of keratoconus. The corneal stroma is soaked with a riboflavin solution before being exposed to ultraviolet-A radiation.

In the current standard CXL, the central corneal epithelium must be debrided to allow the penetration of riboflavin into the cornea with a risk of side effects, such as pain for the first two post-operative days, temporary loss of visual acuity during the first three months, and serious complications such as infection and stromal opacity due to corneal scarring.

Iontophoresis is a non invasive technique in which a weak electric current is used to enhance the penetration of riboflavin into the cornea. The iontophoresis technique could allow intrastromal riboflavin diffusion, while keeping the corneal epithelium on, combining the efficiency of the standard procedure without the side effects of epithelial debridement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Corneal thickness ≥ 400 µm
* Progressive stage 1 to 3 keratoconus (Krumeich classification)

Exclusion Criteria:

* Corneal thickness < 400µm
* Stage 4 keratoconus (Krumeich classification)
* Concomitant corneal disease
* History of corneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
The main outcome parameter is the non-inferiority of iontophoretic CXL compared to standard CXL in progressive keratoconus | Outcome measure is assessed at 1 year.
  Measuring maximum keratometry (K-max) derived from computerized videokeratography.

SECONDARY OUTCOMES:
Comparison of minimum keratometry | 3 months
  Measure assessed by tomographic measurement.

OTHER OUTCOMES:
Comparison of mean keratometry | At 1 year
  Tomographic measurement.
Comparison of postoperative pain and complications during the follow up | Outcome measure is assessed at 1 year and at 3 months
Comparison of visual acuity | Outcome measure is assessed at 1 year and at 3 months
Intraoperative comparison of corneal concentration of riboflavin | Outcome measure is assessed at 1 year and at 3 months
Comparison of depth of treatment | Outcome measure is assessed at 1 year and at 3 months
  By tomographic measurement
Comparison of biomechanical parameters | Outcome measure is assessed at 1 year and at 3 months
  By ORA (Ocular Response Analyzer)
Comparison of corneal thickness | Outcome measure is assessed at 1 year and at 3 months for the tomographic measurement.

CONTACTS AND LOCATIONS:
Overall Officials: François MALECAZE, MD, PhD, Principal Investigator
Locations (1):
- University Hospital Toulouse, Toulouse, Midi-Pyrenees, France

REFERENCES:
- [Background] Krachmer JH, Feder RS, Belin MW. Keratoconus and related noninflammatory corneal thinning disorders. Surv Ophthalmol. 1984 Jan-Feb;28(4):293-322. doi: 10.1016/0039-6257(84)90094-8. PMID 6230745
- [Background] Kennedy RH, Bourne WM, Dyer JA. A 48-year clinical and epidemiologic study of keratoconus. Am J Ophthalmol. 1986 Mar 15;101(3):267-73. doi: 10.1016/0002-9394(86)90817-2. PMID 3513592
- [Background] Rabinowitz YS. Keratoconus. Surv Ophthalmol. 1998 Jan-Feb;42(4):297-319. doi: 10.1016/s0039-6257(97)00119-7. PMID 9493273
- [Background] Zadnik K, Barr JT, Gordon MO, Edrington TB. Biomicroscopic signs and disease severity in keratoconus. Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study Group. Cornea. 1996 Mar;15(2):139-46. doi: 10.1097/00003226-199603000-00006. PMID 8925661
- [Background] AMSLER M. [Classic keratocene and crude keratocene; Unitary arguments]. Ophthalmologica. 1946 Feb-Mar;111(2-3):96-101. doi: 10.1159/000300309. No abstract available. French. PMID 20275788
- [Background] McMahon TT, Edrington TB, Szczotka-Flynn L, Olafsson HE, Davis LJ, Schechtman KB; CLEK Study Group. Longitudinal changes in corneal curvature in keratoconus. Cornea. 2006 Apr;25(3):296-305. doi: 10.1097/01.ico.0000178728.57435.df. PMID 16633030
- [Background] Zadnik K, Steger-May K, Fink BA, Joslin CE, Nichols JJ, Rosenstiel CE, Tyler JA, Yu JA, Raasch TW, Schechtman KB; CLEK Study Group. Collaborative Longitudinal Evaluation of Keratoconus. Between-eye asymmetry in keratoconus. Cornea. 2002 Oct;21(7):671-9. doi: 10.1097/00003226-200210000-00008. PMID 12352084
- [Background] Rabinowitz YS, Nesburn AB, McDonnell PJ. Videokeratography of the fellow eye in unilateral keratoconus. Ophthalmology. 1993 Feb;100(2):181-6. doi: 10.1016/s0161-6420(93)31673-8. PMID 8437824
- [Background] Krumeich JH, Daniel J, Knulle A. Live-epikeratophakia for keratoconus. J Cataract Refract Surg. 1998 Apr;24(4):456-63. doi: 10.1016/s0886-3350(98)80284-8. PMID 9584238
- [Background] Colin J, Malet FJ. Intacs for the correction of keratoconus: two-year follow-up. J Cataract Refract Surg. 2007 Jan;33(1):69-74. doi: 10.1016/j.jcrs.2006.08.057. PMID 17189796
- [Background] Ertan A, Kamburoglu G. Intacs implantation using a femtosecond laser for management of keratoconus: Comparison of 306 cases in different stages. J Cataract Refract Surg. 2008 Sep;34(9):1521-6. doi: 10.1016/j.jcrs.2008.05.028. PMID 18721713
- [Background] Ferrara G, Torquetti L, Ferrara P, Merayo-Lloves J. Intrastromal corneal ring segments: visual outcomes from a large case series. Clin Exp Ophthalmol. 2012 Jul;40(5):433-9. doi: 10.1111/j.1442-9071.2011.02698.x. PMID 21902789
- [Background] Arne JL, Fournie P. [Keratoconus, the most common corneal dystrophy. Can keratoplasty be avoided?]. Bull Acad Natl Med. 2011 Jan;195(1):113-29. French. PMID 22039707
- [Background] Cheng YY, Visser N, Schouten JS, Wijdh RJ, Pels E, van Cleynenbreugel H, Eggink CA, Zaal MJ, Rijneveld WJ, Nuijts RM. Endothelial cell loss and visual outcome of deep anterior lamellar keratoplasty versus penetrating keratoplasty: a randomized multicenter clinical trial. Ophthalmology. 2011 Feb;118(2):302-9. doi: 10.1016/j.ophtha.2010.06.005. Epub 2010 Sep 15. PMID 20832121
- [Background] Epstein RJ, Seedor JA, Dreizen NG, Stulting RD, Waring GO 3rd, Wilson LA, Cavanagh HD. Penetrating keratoplasty for herpes simplex keratitis and keratoconus. Allograft rejection and survival. Ophthalmology. 1987 Aug;94(8):935-44. doi: 10.1016/s0161-6420(87)33356-1. PMID 3309775
- [Background] Kirkness CM, Ficker LA, Steele AD, Rice NS. The success of penetrating keratoplasty for keratoconus. Eye (Lond). 1990;4 ( Pt 5):673-88. doi: 10.1038/eye.1990.95. PMID 2282941
- [Background] The Australian Corneal Graft Registry. 1990 to 1992 report. Aust N Z J Ophthalmol. 1993 May;21(2 Suppl):1-48. PMID 8333942
- [Background] Borderie VM, Boelle PY, Touzeau O, Allouch C, Boutboul S, Laroche L. Predicted long-term outcome of corneal transplantation. Ophthalmology. 2009 Dec;116(12):2354-60. doi: 10.1016/j.ophtha.2009.05.009. Epub 2009 Oct 7. PMID 19815285
- [Background] Spoerl E, Huhle M, Seiler T. Induction of cross-links in corneal tissue. Exp Eye Res. 1998 Jan;66(1):97-103. doi: 10.1006/exer.1997.0410. PMID 9533835
- [Background] Wollensak G, Spoerl E, Seiler T. Stress-strain measurements of human and porcine corneas after riboflavin-ultraviolet-A-induced cross-linking. J Cataract Refract Surg. 2003 Sep;29(9):1780-5. doi: 10.1016/s0886-3350(03)00407-3. PMID 14522301
- [Background] Raiskup-Wolf F, Hoyer A, Spoerl E, Pillunat LE. Collagen crosslinking with riboflavin and ultraviolet-A light in keratoconus: long-term results. J Cataract Refract Surg. 2008 May;34(5):796-801. doi: 10.1016/j.jcrs.2007.12.039. PMID 18471635
- [Background] Wittig-Silva C, Whiting M, Lamoureux E, Lindsay RG, Sullivan LJ, Snibson GR. A randomized controlled trial of corneal collagen cross-linking in progressive keratoconus: preliminary results. J Refract Surg. 2008 Sep;24(7):S720-5. doi: 10.3928/1081597X-20080901-15. PMID 18811118
- [Background] Koller T, Mrochen M, Seiler T. Complication and failure rates after corneal crosslinking. J Cataract Refract Surg. 2009 Aug;35(8):1358-62. doi: 10.1016/j.jcrs.2009.03.035. PMID 19631120
- [Background] Wollensak G, Spoerl E, Seiler T. Riboflavin/ultraviolet-a-induced collagen crosslinking for the treatment of keratoconus. Am J Ophthalmol. 2003 May;135(5):620-7. doi: 10.1016/s0002-9394(02)02220-1. PMID 12719068
- [Background] Caporossi A, Baiocchi S, Mazzotta C, Traversi C, Caporossi T. Parasurgical therapy for keratoconus by riboflavin-ultraviolet type A rays induced cross-linking of corneal collagen: preliminary refractive results in an Italian study. J Cataract Refract Surg. 2006 May;32(5):837-45. doi: 10.1016/j.jcrs.2006.01.091. PMID 16765803
- [Background] Dhawan S, Rao K, Natrajan S. Complications of corneal collagen cross-linking. J Ophthalmol. 2011;2011:869015. doi: 10.1155/2011/869015. Epub 2011 Dec 27. PMID 22254130
- [Background] Mazzotta C, Balestrazzi A, Baiocchi S, Traversi C, Caporossi A. Stromal haze after combined riboflavin-UVA corneal collagen cross-linking in keratoconus: in vivo confocal microscopic evaluation. Clin Exp Ophthalmol. 2007 Aug;35(6):580-2. doi: 10.1111/j.1442-9071.2007.01536.x. PMID 17760642
- [Background] Greenstein SA, Fry KL, Bhatt J, Hersh PS. Natural history of corneal haze after collagen crosslinking for keratoconus and corneal ectasia: Scheimpflug and biomicroscopic analysis. J Cataract Refract Surg. 2010 Dec;36(12):2105-14. doi: 10.1016/j.jcrs.2010.06.067. PMID 21111314
- [Background] Pollhammer M, Cursiefen C. Bacterial keratitis early after corneal crosslinking with riboflavin and ultraviolet-A. J Cataract Refract Surg. 2009 Mar;35(3):588-9. doi: 10.1016/j.jcrs.2008.09.029. PMID 19251154
- [Background] Rama P, Di Matteo F, Matuska S, Paganoni G, Spinelli A. Acanthamoeba keratitis with perforation after corneal crosslinking and bandage contact lens use. J Cataract Refract Surg. 2009 Apr;35(4):788-91. doi: 10.1016/j.jcrs.2008.09.035. PMID 19304108
- [Background] Kymionis GD, Portaliou DM, Bouzoukis DI, Suh LH, Pallikaris AI, Markomanolakis M, Yoo SH. Herpetic keratitis with iritis after corneal crosslinking with riboflavin and ultraviolet A for keratoconus. J Cataract Refract Surg. 2007 Nov;33(11):1982-4. doi: 10.1016/j.jcrs.2007.06.036. PMID 17964410
- [Background] Kymionis GD, Portaliou DM, Pallikaris IG. Additional complications of corneal crosslinking. J Cataract Refract Surg. 2010 Jan;36(1):185; author reply 186. doi: 10.1016/j.jcrs.2009.07.028. No abstract available. PMID 20117734
- [Background] Yuksel N, Bilgihan K, Hondur AM. Herpetic keratitis after corneal collagen cross-linking with riboflavin and ultraviolet-A for progressive keratoconus. Int Ophthalmol. 2011 Dec;31(6):513-5. doi: 10.1007/s10792-011-9489-x. Epub 2011 Dec 3. PMID 22139351
- [Background] Labiris G, Kaloghianni E, Koukoula S, Zissimopoulos A, Kozobolis VP. Corneal melting after collagen cross-linking for keratoconus: a case report. J Med Case Rep. 2011 Apr 16;5:152. doi: 10.1186/1752-1947-5-152. PMID 21496288
- [Background] Ghanem RC, Netto MV, Ghanem VC, Santhiago MR, Wilson SE. Peripheral sterile corneal ring infiltrate after riboflavin-UVA collagen cross-linking in keratoconus. Cornea. 2012 Jun;31(6):702-5. doi: 10.1097/ICO.0b013e318226da53. PMID 22378115
- [Background] Vinciguerra P, Albe E, Romano MR, Sabato L, Trazza S. Stromal opacity after cross-linking. J Refract Surg. 2012 Mar;28(3):165. doi: 10.3928/1081597X-20120301-04. No abstract available. PMID 22373029
- [Background] Rodriguez-Ausin P, Gutierrez-Ortega R, Arance-Gil A, Romero-Jimenez M, Fuentes-Paez G. Keratopathy after cross-linking for keratoconus. Cornea. 2011 Sep;30(9):1051-3. doi: 10.1097/ICO.0b013e3182096789. PMID 21464703
- [Background] Lim LS, Beuerman R, Lim L, Tan DT. Late-onset deep stromal scarring after riboflavin-UV-A corneal collagen cross-linking for mild keratoconus. Arch Ophthalmol. 2011 Mar;129(3):360-2. doi: 10.1001/archophthalmol.2011.23. No abstract available. PMID 21402996
- [Background] Kymionis GD, Portaliou DM, Diakonis VF, Kounis GA, Panagopoulou SI, Grentzelos MA. Corneal collagen cross-linking with riboflavin and ultraviolet-A irradiation in patients with thin corneas. Am J Ophthalmol. 2012 Jan;153(1):24-8. doi: 10.1016/j.ajo.2011.05.036. Epub 2011 Sep 8. PMID 21861976
- [Background] Zhang ZY. Corneal endothelial damage in the relatively thin cornea after collagen cross-linking treatment. Cornea. 2012 Aug;31(8):967; author reply 967-8. doi: 10.1097/ICO.0b013e31824d4254. No abstract available. PMID 22668580
- [Background] Spoerl E, Hoyer A, Pillunat LE, Raiskup F. Corneal cross-linking and safety issues. Open Ophthalmol J. 2011 Feb 11;5:14-6. doi: 10.2174/1874364101105010014. PMID 21399770
- [Background] Ghanem VC, Ghanem RC, de Oliveira R. Postoperative pain after corneal collagen cross-linking. Cornea. 2013 Jan;32(1):20-4. doi: 10.1097/ICO.0b013e31824d6fe3. PMID 22547128
- [Background] Baiocchi S, Mazzotta C, Cerretani D, Caporossi T, Caporossi A. Corneal crosslinking: riboflavin concentration in corneal stroma exposed with and without epithelium. J Cataract Refract Surg. 2009 May;35(5):893-9. doi: 10.1016/j.jcrs.2009.01.009. PMID 19393890
- [Background] Al-Aqaba M, Calienno R, Fares U, Otri AM, Mastropasqua L, Nubile M, Dua HS. The effect of standard and transepithelial ultraviolet collagen cross-linking on human corneal nerves: an ex vivo study. Am J Ophthalmol. 2012 Feb;153(2):258-266.e2. doi: 10.1016/j.ajo.2011.07.006. Epub 2011 Sep 17. PMID 21930257
- [Background] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T, Paradiso AL. Transepithelial corneal collagen crosslinking for keratoconus: qualitative investigation by in vivo HRT II confocal analysis. Eur J Ophthalmol. 2012;22 Suppl 7:S81-8. doi: 10.5301/ejo.5000125. PMID 22344471
- [Background] Boxer Wachler BS, Pinelli R, Ertan A, Chan CC. Safety and efficacy of transepithelial crosslinking (C3-R/CXL). J Cataract Refract Surg. 2010 Jan;36(1):186-8; author reply 188-9. doi: 10.1016/j.jcrs.2009.08.019. No abstract available. PMID 20117737
- [Background] Filippello M, Stagni E, O'Brart D. Transepithelial corneal collagen crosslinking: bilateral study. J Cataract Refract Surg. 2012 Feb;38(2):283-91. doi: 10.1016/j.jcrs.2011.08.030. Epub 2011 Nov 21. PMID 22104644
- [Background] Leccisotti A, Islam T. Transepithelial corneal collagen cross-linking in keratoconus. J Refract Surg. 2010 Dec;26(12):942-8. doi: 10.3928/1081597X-20100212-09. Epub 2010 Feb 15. PMID 20166621
- [Background] Koppen C, Wouters K, Mathysen D, Rozema J, Tassignon MJ. Refractive and topographic results of benzalkonium chloride-assisted transepithelial crosslinking. J Cataract Refract Surg. 2012 Jun;38(6):1000-5. doi: 10.1016/j.jcrs.2012.01.024. PMID 22624899
- [Background] Zhang ZY, Zhang XR. Efficacy and safety of transepithelial corneal collagen crosslinking. J Cataract Refract Surg. 2012 Jul;38(7):1304; author reply 1304-5. doi: 10.1016/j.jcrs.2012.05.012. No abstract available. PMID 22727312
- [Background] Costello CT, Jeske AH. Iontophoresis: applications in transdermal medication delivery. Phys Ther. 1995 Jun;75(6):554-63. doi: 10.1093/ptj/75.6.554. PMID 7770500
- [Background] von Sallmann L. Iontophoretic introduction of atropine and scopolamine into the rabbit eye. Arch Ophthalmol 1943;29:711-9.
- [Background] Jones RF, Maurice DM. New methods of measuring the rate of aqueous flow in man with fluorescein. Exp Eye Res. 1966 Jul;5(3):208-20. doi: 10.1016/s0014-4835(66)80009-x. No abstract available. PMID 5914653
- [Background] Hughes L, Maurice DM. A fresh look at iontophoresis. Arch Ophthalmol. 1984 Dec;102(12):1825-9. doi: 10.1001/archopht.1984.01040031483028. PMID 6508622
- [Background] Lam TT, Edward DP, Zhu XA, Tso MO. Transscleral iontophoresis of dexamethasone. Arch Ophthalmol. 1989 Sep;107(9):1368-71. doi: 10.1001/archopht.1989.01070020438050. PMID 2783069
- [Background] Behar-Cohen F, El Aouni A, Le Rouic JF, Parel JM, Renard G, Chauvaud D. [Iontophoresis: past and future]. J Fr Ophtalmol. 2001 Mar;24(3):319-27. No abstract available. French. PMID 11285450
- [Background] Behar-Cohen FF, Savoldelli M, Parel JM, Goureau O, Thillaye-Goldenberg B, Courtois Y, Pouliquen Y, de Kozak Y. Reduction of corneal edema in endotoxin-induced uveitis after application of L-NAME as nitric oxide synthase inhibitor in rats by iontophoresis. Invest Ophthalmol Vis Sci. 1998 May;39(6):897-904. PMID 9579469
- [Background] Behar-Cohen FF, Parel JM, Pouliquen Y, Thillaye-Goldenberg B, Goureau O, Heydolph S, Courtois Y, De Kozak Y. Iontophoresis of dexamethasone in the treatment of endotoxin-induced-uveitis in rats. Exp Eye Res. 1997 Oct;65(4):533-45. doi: 10.1006/exer.1997.0364. PMID 9464186
- [Background] Chauvaud D, Behar-Cohen F, Parel JM, Renard G. Transscleral iontophoresis of corticosteroids: Phase II Clinical Trial. ARVO Invest Ophthalmol Vis Sci 2000;41:S79.
- [Background] Yoo SH, Dursun D, Dubovy S, Miller D, Alfonso E, Forster RK, Behar-Cohen F, Parel JM. Lontophoresis for the treatment of paecilomyces keratitis. Cornea. 2002 Jan;21(1):131-2. doi: 10.1097/00003226-200201000-00029. No abstract available. PMID 11805526
- [Background] Parkinson TM, Ferguson E, Febbraro S, Bakhtyari A, King M, Mundasad M. Tolerance of ocular iontophoresis in healthy volunteers. J Ocul Pharmacol Ther. 2003 Apr;19(2):145-51. doi: 10.1089/108076803321637672. PMID 12804059
- [Background] Horwath-Winter J, Schmut O, Haller-Schober EM, Gruber A, Rieger G. Iodide iontophoresis as a treatment for dry eye syndrome. Br J Ophthalmol. 2005 Jan;89(1):40-4. doi: 10.1136/bjo.2004.048314. PMID 15615744
- [Background] Behar-Cohen FF, El Aouni A, Gautier S, David G, Davis J, Chapon P, Parel JM. Transscleral Coulomb-controlled iontophoresis of methylprednisolone into the rabbit eye: influence of duration of treatment, current intensity and drug concentration on ocular tissue and fluid levels. Exp Eye Res. 2002 Jan;74(1):51-9. doi: 10.1006/exer.2001.1098. PMID 11878818
- [Background] Eljarrat-Binstock E, Orucov F, Frucht-Pery J, Pe'er J, Domb AJ. Methylprednisolone delivery to the back of the eye using hydrogel iontophoresis. J Ocul Pharmacol Ther. 2008 Jun;24(3):344-50. doi: 10.1089/jop.2007.0097. PMID 18476804
- [Background] Patane MA, Cohen A, From S, Torkildsen G, Welch D, Ousler GW 3rd. Ocular iontophoresis of EGP-437 (dexamethasone phosphate) in dry eye patients: results of a randomized clinical trial. Clin Ophthalmol. 2011;5:633-43. doi: 10.2147/OPTH.S19349. Epub 2011 May 15. PMID 21629568
- [Background] Cohen AE, Assang C, Patane MA, From S, Korenfeld M; Avion Study Investigators. Evaluation of dexamethasone phosphate delivered by ocular iontophoresis for treating noninfectious anterior uveitis. Ophthalmology. 2012 Jan;119(1):66-73. doi: 10.1016/j.ophtha.2011.07.006. Epub 2011 Nov 23. PMID 22115712
- [Background] Wollensak G, Spoerl E, Wilsch M, Seiler T. Endothelial cell damage after riboflavin-ultraviolet-A treatment in the rabbit. J Cataract Refract Surg. 2003 Sep;29(9):1786-90. doi: 10.1016/s0886-3350(03)00343-2. PMID 14522302
- [Background] Spoerl E, Seiler T. Techniques for stiffening the cornea. J Refract Surg. 1999 Nov-Dec;15(6):711-3. doi: 10.3928/1081-597X-19991101-21. PMID 10590015
- [Background] Chien YW, Banga AK. Iontophoretic (transdermal) delivery of drugs: overview of historical development. J Pharm Sci. 1989 May;78(5):353-4. doi: 10.1002/jps.2600780502. No abstract available. PMID 2664122
- [Background] Reinhart WJ, Musch DC, Jacobs DS, Lee WB, Kaufman SC, Shtein RM. Deep anterior lamellar keratoplasty as an alternative to penetrating keratoplasty a report by the american academy of ophthalmology. Ophthalmology. 2011 Jan;118(1):209-18. doi: 10.1016/j.ophtha.2010.11.002. PMID 21199711
- [Background] Caporossi A, Mazzotta C, Baiocchi S, Caporossi T. Long-term results of riboflavin ultraviolet a corneal collagen cross-linking for keratoconus in Italy: the Siena eye cross study. Am J Ophthalmol. 2010 Apr;149(4):585-93. doi: 10.1016/j.ajo.2009.10.021. Epub 2010 Feb 6. PMID 20138607
- [Background] Asri D, Touboul D, Fournie P, Malet F, Garra C, Gallois A, Malecaze F, Colin J. Corneal collagen crosslinking in progressive keratoconus: multicenter results from the French National Reference Center for Keratoconus. J Cataract Refract Surg. 2011 Dec;37(12):2137-43. doi: 10.1016/j.jcrs.2011.08.026. PMID 22108109
- [Background] Vimalin J, Gupta N, Jambulingam M, Padmanabhan P, Madhavan HN. The effect of riboflavin-UV-A treatment on corneal limbal epithelial cells--a study on human cadaver eyes. Cornea. 2012 Sep;31(9):1052-9. doi: 10.1097/ICO.0b013e3182498902. PMID 22673851
- [Result] Touboul D, Robinet-Perrin A, Fournie P, Malecaze F. [Efficacy of corneal cross-linking for the treatment of keratoconus]. J Fr Ophtalmol. 2016 Mar;39(3):308-14. doi: 10.1016/j.jfo.2015.12.002. Epub 2016 Mar 16. French. PMID 26995077